CLINICAL TRIAL: NCT07306208
Title: The Effect of Sexual Health Education Provided Using the Flipped Classroom Method on University Students' Sexual Health Literacy Levels: A Randomised Controlled Trial
Brief Title: Flipped Classroom Sexual Health Education Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Hafize Dağ Tüzmen, Principal Investigator, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SHL KARATAY
Record Dates: First submitted 2025-12-12; First posted 2025-12-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Sexual Health; Health Literacy; Health Education; Flipped Classroom Model in Teaching; Randomized Controlled Trial
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flipped Classroom (Experimental): The intervention group received a structured sexual health education program based on a flipped classroom approach. The program was supported by videos, reading materials, and digital presentations during the pre-learning phase; synchronous sessions utilized active learning methods such as case discussions, role-playing, and group activities. The training was conducted weekly for 10 weeks as 90-minute online sessions.
  Interventions: Behavioral: Flipped learning
- CONTROL (No Intervention): Students in the control group received the same sexual health curriculum using traditional teaching methods. Instruction was delivered through question-and-answer sessions and synchronous online classes; 10 sessions, each lasting 90 minutes, were matched to the session durations of the intervention group.

INTERVENTIONS:
Behavioral: Flipped learning — Students in this group will be offered a sexual health education programme developed in line with structured learning objectives and organised according to the flipped learning approach. The training will be supported by video lectures, reading materials and digital presentations during the pre-learning phase, while active learning strategies such as case discussions, role-playing and group activities will be implemented in synchronous sessions. The training will be conducted over a total of 10 weeks, with 90-minute online sessions held once a week. All content will be prepared by researchers and subject matter experts, and content validity will be ensured.
  Arms: Flipped Classroom

SUMMARY:
Sexual health is an integral component of individuals' physical, emotional, mental, and social well-being. Lack of knowledge and cultural taboos negatively affect individuals' ability to make informed decisions and adopt protective behaviors. Therefore, effective sexual health education is of great importance. The flipped learning method, a student-centered approach, promotes active participation and long-term learning. This study aimed to examine the effect of sexual health education delivered through the flipped learning method on university students' sexual health knowledge levels and sexual health literacy.

DETAILED DESCRIPTION:
This study is a randomized controlled experimental research designed using quantitative methods and was conducted between September and November 2025 at two private universities in Konya and Mersin. The study included individuals aged 18 and over who were nursing or midwifery students, had access to online education, and had not previously received structured sexual health education. Those who did not attend more than 20% of the training, did not complete the assessment tools, had previously received formal sexual health education, and withdrew from the study without justification were excluded.

The intervention group received structured sexual health education based on a flipped classroom approach; weekly 90-minute online sessions were conducted for 10 weeks, including pre-learning materials and active learning methods. The control group received the same curriculum using traditional teaching methods, matched to the intervention group in terms of duration and number of sessions.

Data were collected using the Personal Information Form (PIF) and the Sexual Health Literacy Scale (SHLS).

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Being enrolled in a health-related department at a university
* Having internet access and the technical equipment required to follow online training sessions
* Not having previously participated in a structured sexual health education program with similar content

Exclusion Criteria:

* Studying in health departments where the instructors of the training are teaching
* Attending less than 80% of the training sessions (missing 3 or more sessions)
* Failing to complete the assessment tools without a valid excuse during the study
* Having previously received formal sexual health education
* Voluntarily withdrawing from the study without providing a reason

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2025-11-02 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2026-01-19 (Actual)

PRIMARY OUTCOMES:
Sexual Health Literacy | Baseline (pretest), Week 5 (follow-up test), Week 10 (posttest)
  It will be measured using the Sexual Health Literacy Scale.The minimum score obtainable on the scale is 17, while the maximum score is 85. An increase in scores indicates that the individual has a high level of sexual health literacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Kto Karatay University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data supporting the findings of this study are available from the corresponding author upon reasonable request.